CLINICAL TRIAL: NCT03240458
Title: Screening For Diabetic Macular Edema Among Diabetic Patients In Assiut University Hospital Using Optical Coherence Tomography
Brief Title: Screening For Diabetic Macular Edema Among Diabetic Patients Using Optical Coherence Tomography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara maksoud, principle investgator, Assiut University
Other Study IDs: DMEDP
Record Dates: First submitted 2017-07-13; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-07

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Optical Coherence Tomography — an objective non-invasive method for high-resolution cross-sectional imaging of the retina

SUMMARY:
Diabetic macular edema is one of the major causes of visual impairment in diabetic retinopathy patients especially in the working age group. The problem is likely to increase in the future with statistics showing a growing number of the diabetic population especially in the Middle East . .

DETAILED DESCRIPTION:
The worldwide prevalence of diabetic macular edema was reported as 6.81% among patients with diabetes. Other research reported that the 10-year incidence of diabetic macular edema was 14% in individuals with type 2 diabetes, and progression to diabetic macular edema occurred in 29% of individuals with type 1 diabetes over 25 years if left untreated . Although diabetic macular edema resolves spontaneously in about 33% to 35% of patients, it tends to be chronic in most patients..Diabetic macular edema can occur at any stage of diabetic retinopathy . The symptoms of diabetic macular range from slight visual blurring to complete blindness if left untreated . Optical coherence tomography is an objective non-invasive method for high-resolution cross-sectional imaging of the retina .

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1or type 2 Diabetes Mellitus.
* Fundus examination and optical coherence tomography can be done with no significant hazy media

Exclusion Criteria:

1. Previous ocular surgery (e.g. vitreo-retinal surgery, glaucoma surgery).
2. Presence of co-existing retinal or choroidal disease (e.g. high myopia, retinitis pigmentosa and Age-related macular degeneration)
3. Other associated ocular conditions (ex. glaucoma & corneal opacity & iritis).
4. Previous history of trauma.
5. Pregnancy induced diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-08-10 (Estimated); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
The prevalence of diabetic macular edema in diabetic patients | 5 minutes
  The prevalence of diabetic macular edema in diabetic patients using optical coherence tomography .

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Sayed, Lecturer, Study Chair — Assiut University

REFERENCES:
- [Background] Studnicka J. [The diabetic macular edema--new possibilities of the treatment]. Cesk Slov Oftalmol. 2012 May;68(2):61-3. Czech. PMID 22913868
- [Background] Klein R, Klein BE, Moss SE, Cruickshanks KJ. The Wisconsin Epidemiologic Study of Diabetic Retinopathy. XV. The long-term incidence of macular edema. Ophthalmology. 1995 Jan;102(1):7-16. doi: 10.1016/s0161-6420(95)31052-4. PMID 7831044
- [Background] Klein R, Knudtson MD, Lee KE, Gangnon R, Klein BE. The Wisconsin Epidemiologic Study of Diabetic Retinopathy: XXII the twenty-five-year progression of retinopathy in persons with type 1 diabetes. Ophthalmology. 2008 Nov;115(11):1859-68. doi: 10.1016/j.ophtha.2008.08.023. PMID 19068374
- [Background] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Background] Zhang J, Ma J, Zhou N, Zhang B, An J. Insulin use and risk of diabetic macular edema in diabetes mellitus: a systemic review and meta-analysis of observational studies. Med Sci Monit. 2015 Mar 30;21:929-36. doi: 10.12659/MSM.892056. PMID 25816765
- [Background] Romero-Aroca P, Reyes-Torres J, Baget-Bernaldiz M, Blasco-Sune C. Laser treatment for diabetic macular edema in the 21st century. Curr Diabetes Rev. 2014 Mar;10(2):100-12. doi: 10.2174/1573399810666140402123026. PMID 24852439
- [Background] Das A, McGuire PG, Rangasamy S. Diabetic Macular Edema: Pathophysiology and Novel Therapeutic Targets. Ophthalmology. 2015 Jul;122(7):1375-94. doi: 10.1016/j.ophtha.2015.03.024. Epub 2015 Apr 30. PMID 25935789
- [Background] Varma R, Bressler NM, Doan QV, Gleeson M, Danese M, Bower JK, Selvin E, Dolan C, Fine J, Colman S, Turpcu A. Prevalence of and risk factors for diabetic macular edema in the United States. JAMA Ophthalmol. 2014 Nov;132(11):1334-40. doi: 10.1001/jamaophthalmol.2014.2854. PMID 25125075